CLINICAL TRIAL: NCT03172871
Title: A Multicenter, Randomized, Double-blind, Active-Controlled Study to Evaluate the Efficacy and Safety of Aripiprazole Intramuscular Depot in the Acute Treatment of Adults With Schizophrenia
Brief Title: Aripiprazole IM Depot in the Acute Treatment of Adults With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-403-00048
Record Dates: First submitted 2017-05-11; First posted 2017-06-01 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Aripiprazole Intramuscular Depot; Acute treatment
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole IM Depot (Experimental): Aripiprazole IM depot group (Aripiprazole IM Depot):
  The first 2 weeks of the acute treatment phase IM Injection 400 mg every 4 weeks + Aripiprazole tablets 10-20 mg per day After the first two weeks of the acute treatment phase IM Injection 400/300 mg every 4 weeks + placebo（tablets）(once a day)
  Interventions: Drug: Aripiprazole IM Depot; Drug: Aripiprazole tablet
- Aripiprazole tablet (Active Comparator): Oral aripiprazole group (Aripiprazole tablet):
  The first 2 weeks of the acute treatment phase Placebo (Injection) every 4 weeks + Aripiprazole tablets 10-20 mg per day After the first two weeks of the acute treatment phase Placebo (Injection) every 4 weeks + Aripiprazole tablets 10-20 mg per day
  Interventions: Drug: Aripiprazole IM Depot; Drug: Aripiprazole tablet

INTERVENTIONS:
Drug: Aripiprazole IM Depot — Aripiprazole IM depot 400 mg/300 mg (when not tolerated)
  Other Names: Aripiprazole Intramuscular Depot
Drug: Aripiprazole tablet — Oral aripiprazole tablets 10 to 20 mg daily
  Other Names: Aripiprazole TAB

SUMMARY:
This is a phase 3, multicenter, randomized, active-controlled trial to assess the efficacy and safety of aripiprazole Intramuscular Depot in the acute treatment of adults with schizophrenia. The trial will include a 13-day screening phase and a 12-week acute treatment phase with a 14(±2)-day safety follow-up.

DETAILED DESCRIPTION:
Screening Phase: The screening phase will begin when informed consent is signed and be a maximum of 13 days. The investigators will assess the subjects who meet all eligibility criteria and collect the characteristic information of the subjects, such as demographic, medical history, etc. If subjects have been exposed to aripiprazole in the past (ie, tolerability has been established), then subjects will enter a washout period for 3～7 days from prior antipsychotic medications and other prohibited concomitant medications. If the investigator may reasonably verify that subject has been off antipsychotics for at least 3～7 days and has a history of tolerating aripiprazole, then the subject may have a screening phase of < 7 days as long as the subject has had at least a 3～7-day washout phase from other antipsychotic medications. Subjects are required to be hospitalized during the entire screening phase.

12-week Acute Treatment Phase: At baseline, eligible subjects will be randomized in a 1:1 ratio to either aripiprazole IM depot or aripiprazole tablet. For 14 days beginning with the first injection, subjects randomized aripiprazole IM depot will receive concomitant oral aripiprazole and subjects randomized to aripiprazole tablet will receive 12 weeks concomitant injection placebo.

Safety Follow-up Phase: All subjects will be followed-up for safety via telephone contact 14(±2) days after the last trial visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent form by subjects and subject's legal guardian or legally acceptable representative.
2. The subjects and subject's legal guardian or legally acceptable representative have the ability to understand the nature of the trial, agree to comply with the prescribed medication and dosage regimens, complete the schedule visit, report the adverse event and concomitant medication to investigator, and to be reliably rated on psychiatrically scales.
3. Male and female subjects 18 to 65 years of age, at the time of informed consent.
4. Subjects with a diagnosis of schizophrenia as defined by DSM-IV-TR criteria and confirmed by the MINI for Schizophrenia and Psychotic Disorders Studies.
5. Subjects with a stable living environment when not in hospital, as demonstrated by the ability to provide contact information for themselves and/or family/friend(s)/caregiver(s).
6. Subjects who are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by meeting BOTH of the following at screening and baseline:

   * Currently experiencing an acute exacerbation of psychotic symptoms accompanied by significant deterioration in the subject's clinical and/or functional status from their baseline clinical presentation with a Positive and Negative Syndrome Scale (PANSS) Total Score≥ 70 AND
   * Specific psychotic symptoms on the PANSS as measured by a score of > 4 on at least two of the following items (possible scores of 1 to 7 for each item) Conceptual disorganization (P2) Hallucinatory behavior (P3) Suspiciousness/persecution (P6) Unusual thought content (G9)
7. According to the investigator's opinion, subjects who have received antipsychotic treatment (except clozapine) with good response. (this criteria only applicable for the schizophrenia recurrence subject).
8. Subjects willing to discontinue all prohibited psychotropic medications to meet protocol requirements prior to and during the trial period.

Exclusion Criteria

1. Woman and men subjects with Child-bear potential, unwilling or unable to take effective contraception within 1 year after signing informed consent form.
2. Women who are pregnant or breastfeeding.
3. Subjects with improvement of ≥ 30% in total PANSS score between the screening and baseline assessments.
4. Subjects hospitalized for ≥ 30 days out of the last 90 days prior to screening visit. Subjects who have been hospitalized > 5 days for the current acute episode at the time of the screening visit (ie, signing the informed consent).
5. Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history of failure to respond to 2 adequate trials with different antipsychotic medications with a minimum of 6 weeks at clinically efficacious tolerated doses. Subjects who have a history of response to clozapine treatment only.
6. Subjects with a current Axis I (DSM-IV-TR) diagnosis other than schizophrenia including, but not limited to:

   Delirium, dementia, amnesic or other cognitive disorder MDD, schizoaffective disorder, or other psychotic disorder Bipolar I or II disorder Eating disorder (including anorexia nervosa or bulimia) Obsessive compulsive disorder Panic disorder Post-traumatic stress disorder
7. Subjects with a current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.
8. Subjects experiencing acute depressive symptoms within the past 30 days, according to the investigator's opinion, that require treatment with an antidepressant.
9. Subjects who present a serious risk of suicide, as follows:

   Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 6 months OR Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Subjects who, in the opinion of the investigator, present a serious risk of suicide.
10. Subjects with clinically significant tardive dyskinesia, as determined by a score of ≥ 3 on Item 8 of the AIMS at the screening visit.
11. Subjects with a score of 5 (severe akathisia) on the BARS global clinical assessment of akathisia at screening or baseline.
12. Subjects who have met DSM-IV-TR criteria for substance abuse with the past 3 months prior to screening or dependence within the past 6 months; including alcohol and benzodiazepines, but excluding caffeine and nicotine.
13. Subjects who have a history or severe organic disease of vital organs (including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease ).
14. Subjects with insulin-dependent diabetes mellitus or non-insulin-dependent diabetes mellitus are excluded if their illness is unstable as evidenced by any of the following:

    HbA1c≥ 7.0% OR Screening glucose ≥ 125 mg/dL or ≥ 6.94 mmol/L (fasting) or ≥ 200 mg/dL or ≥ 11.1 mmol/L (nonfasting). If the fasting or nonfasting screening glucose is greater than the above values, subjects must be retested in a fasted state and the retest value must be ≥125 mg/dL or ≥ 6.94 mmol/L, OR Subject's diabetes is newly diagnosed during screening for the trial.
15. Subjects with uncontrolled hypertension (DBP > 95 mmHg in any position) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in SBP and/or a decrease of ≥ 20 mmHg in DBP after at least 3 minutes standing compared to the previous supine blood pressure, OR development of symptoms.
16. Subjects with known ischemic heart disease or history of myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery.
17. Subjects with epilepsy or a history of seizures, except for a single seizure episode, for instance childhood febrile seizure, post traumatic, or alcohol withdrawal.
18. The following laboratory test and ECG results are exclusionary 1) Platelets ≤ 75 000/mm3 OR ≤ 75 × 109 /L 2) Hemoglobin ≤9 g/dL OR ≤90 g/L 3) Neutrophils, absolute ≤ 1 000/mm3 OR ≤ 1 × 109 /L 4) AST > 3 × ULN OR ALT > 3 × ULN 5) CPK > 3 × ULN 6) Creatinine≥ 2 mg/dL OR ≥ 176.8 µmol/L 7) HbA1c ≥ 7.0% 8) QTc ≥450 msec (male) OR QTc ≥470 msec (female)
19. BMI> 40 kg/m2 (morbid obesity)at screening
20. Prohibited concomitant medications used prior to randomization or anticipated need for such medications during the trial, including, but not limited to, the following:

    Medication Required Washout Antipsychotics Oral (or IR IM) aripiprazole 3∼7 days Other oral (or IR IM) antipsychotics 3∼7 days Depot or long-acting injectable antipsychotics One full cycle plus 14 days (length of 1 cycle plus 14 days base on the prescribing label） Antidepressants Fluoxetine or Symbyax® 28 days Venlafaxina and desvenlafaxine 3 days All other andtidepressants including MAOIs 3∼7 days Mood stabilizers(ie，lithium and/or anticonvulsants） 3∼7 days Psychostimulants 3∼7 days Varenicine 3∼7 days Benzodiazepines Lorazepam, oxazepam, diazepam, or clonazepam (rescue therapy during washout) 12 hours before scales Other benzodiazepines 3∼7 days CYP3A4 inhibitors and inducers and CYP2D6 inhibitors 3∼7 days
21. Subjects who received electroconvulsive therapy within 60 days of screening.
22. Subjects who previously enrolled in any prior aripiprazole IM depot clinical trial regardless if they received an injection of investigational medicinal product (IMP) or not.
23. Subjects with a history of neuroleptic malignant syndrome (NMS)
24. Subjects with a history of true allergic response (ie, not intolerance) to more than 1 class of medications.
25. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness must not be enrolled into this trial.
26. Subjects who anticipated any other clinical trial within 3 months prior to the informed consent form.
27. Any subject who, in the opinion of the investigator, should not participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint(10th week)in PANSS Total Score. | 1st,2nd,4th,6th,8th,10th,12th week
  The primary efficacy outcome variable is mean change from baseline to endpoint (Week 10) in PANSS Total Score. The objective of the primary analysis is to compare the efficacy of aripiprazole IM depot (400 mg or 300 mg) with that of placebo with regard to mean change from baseline to endpoint (Week 10) in PANSS Total Score.

CONTACTS AND LOCATIONS:
Overall Officials: Patyman Juma, Study Director — Otsuka Beijing Research Institute
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao L, Zhao Q, Li AN, Sun J, Wu B, Wang L, Zhang H, Zhang R, Li K, Xu X, Liu T, Zhang W, Xie S, Xu X, Tan Y, Zhang K, Zhang H, Guan N, Xian M, Uki M, Wang G. Efficacy and safety of aripiprazole once-monthly versus oral aripiprazole in Chinese patients with acute schizophrenia: a multicenter, randomized, double-blind, non-inferiority study. Psychopharmacology (Berl). 2022 Jan;239(1):243-251. doi: 10.1007/s00213-021-06044-x. Epub 2022 Jan 6. PMID 34989824